CLINICAL TRIAL: NCT06653322
Title: A Multi-centered，Randomized，Double-blind，Placebo-controlled Study to Evaluate the Efficacy and Safety of SHR-1703 in Eosinophilic Asthma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1703-302
Record Dates: First submitted 2024-10-20; First posted 2024-10-22 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Asthma With Eosinophilic Phenotype

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects receiving SHR-1703 dose 1 (Experimental)
  Interventions: Drug: HR-1703
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HR-1703 — HR-1703 will be administered by SC injection.
  Arms: Subjects receiving SHR-1703 dose 1
Drug: Placebo — Matching Placebo will be administered by the SC injection.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the Pharmacodynamic, Efficacy and Safety of SHR-1703 in Asthma Patients with Eosinophil Phenotype

ELIGIBILITY:
Inclusion Criteria:

1. At least 12 years of age
2. A minimum weight of 40kg
3. A medical history of at least 1 year that meets the diagnosis of asthma;
4. Current treatment with medium- or high- doses of ICS for at least 6 months and using steadily at least 3 months
5. Current treatment with an additional controller medication, besides ICS, for at least 3 months and using steadily at least 1 month
6. Absolute count of blood eosinophils suggests eosinophilic asthma
7. During the screening period and baseline, pre- BD FEV1% < 80%
8. During the screening period and baseline, ACQ-6 score indicates asthma poor control
9. History of severe asthma exacerbation within the past 12 months prior to screening
10. Good compliance with eDiary completion
11. Take efficient contraceptive measures
12. Voluntarily sign the informed consent form to participate in this study

Exclusion Criteria:

1. With other condition that could lead to elevated eosinophils
2. With Clinically significant pulmonary diseases
3. With existing immunodeficiency disease
4. With other clinically significant diseases that may affect lung function
5. With uncontrolled severe cardiovascular and cerebrovascular diseases
6. With uncontrolled hypertension and/or diabetes
7. With exacerbation, allergic rhinitis or sinusitis attacks, or clinical significant infection requiring intervention during 4 weeks prior to randomization
8. Recent major surgeries or surgical plans during the study period, or treatment measures that investigators believe may affect subject evaluation
9. Existing parasitic infections
10. Diagnosed as malignant tumor within the first 5 years of randomization
11. Significant abnormalities in screening period or baseline laboratory tests
12. Screening period or baseline ECG QTc prolongation
13. Prohibited drugs using during the pre randomization period
14. Participated in other clinical trials within 30 days prior to screening and used research drugs containing active ingredients, or was still within 5 half lives of the research drug at the time of screening
15. Smoking or quitting smoking for less than 6 months during screening, or previous smoking history ≥ 10 pack years
16. History of drug use, alcoholism, or substance abuse within the past year prior to screening
17. Allergic or intolerant to IL-5 monoclonal antibodies or other biological agents
18. Pregnant or lactating subjects
19. Other reasons why the researcher deemed it unsuitable for conducting this experiment

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Annualised asthma exacerbation rate，about 48weeks | about 48weeks

SECONDARY OUTCOMES:
Mean number of days with oral corticosteroids taken for exacerbation，about 48weeks | about 48weeks
Frequency of exacerbations requiring hospitalisation，about 48weeks | about 48weeks
Time to first exacerbation requiring hospitalisation，about 48weeks | about 48weeks
Mean change from baseline in clinic pre- and post-BD FEV1，about 64 weeks | about 64 weeks
Mean change from baseline in clinic pre- and post-BD FEV1%，about 64weeks | about 64weeks
Mean change from baseline in clinic pre- and post-BD FVC，about 64 weeks | about 64 weeks
Mean change from baseline in clinic pre- and post-BD PEF，about 64 weeks | about 64 weeks
Mean change from baseline in FeNO，about 64weeks | about 64weeks
Mean change from baseline in asthma control questionnaire (ACQ-6) score，about 64 weeks | about 64 weeks
Mean change from baseline in ASTHMA QUALITY OF LIFE QUESTIONNAIRES (AQLQ) score，about 64weeks | about 64weeks
Mean change from baseline in Asthma symptom score at week 12/24/36/48/60，about 64weeks | at week 12/24/36/48/60，about 64weeks
Mean change from baseline in daily rescue medication use at week 12/24/36/48/60，about 64weeks | at week 12/24/36/48/60，about 64weeks
Mean change from baseline in awakening at night due to asthma symptoms requiring rescue medication use at week 12/24/36/48/60，about 64weeks | at week 12/24/36/48/60，about 64weeks
Mean change from baseline in morning and evening PEF at week 12/24/36/48/60，about 64weeks | at week 12/24/36/48/60，about 64weeks
Mean change from baseline in IgE，about 64weeks | about 64weeks
Adverse events，about 64weeks | about 64weeks

CONTACTS AND LOCATIONS:
Locations (1):
- West China School of Medicine West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided